CLINICAL TRIAL: NCT02547441
Title: A Phase 3, Randomized, Vehicle-Controlled, Double-Blind, Multicenter Study to Evaluate the Safety and Efficacy of a Once-Daily CLS001 Topical Gel Versus Vehicle Administered for 12 Weeks to Subjects With Papulopustular Rosacea With an Open-Label Safety Extension
Brief Title: Study to Evaluate the Safety and Efficacy of a Once-Daily CLS001 Topical Gel Versus Vehicle
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLS001-CO-PR-004
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Results first posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Omiganan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): CLS001 (Omiganan) gel applied once daily
  Interventions: Drug: CLS001 (Omiganan)
- Vehicle Gel (Placebo Comparator): Vehicle gel applied once daily
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: CLS001 (Omiganan) — Topical gel
  Arms: Treatment
Drug: Vehicle — Vehicle Gel
  Arms: Vehicle Gel

SUMMARY:
This study evaluates the safety and efficacy of once-daily application of CLS001 topical gel compared to vehicle gel in subjects with severe papulopustular rosacea.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male and non-pregnant female subjects, 18 years of age or older.
2. A diagnosis of papulopustular rosacea with ≥30 inflammatory facial lesions at Baseline. Subjects must have no more than 2 nodular lesions, at Baseline.
3. Subjects with the presence of telangiectasia at Baseline.
4. Subjects with an erythema score of at least 2 on the Investigator Assessment of Erythema scale at Baseline.
5. Subjects with severe rosacea on the Investigators Global Assessment scale at Baseline.

Exclusion Criteria:

1. Subjects with steroid rosacea or subtype 3 (phymatous rosacea).
2. Subjects with nodular rosacea.
3. Standard exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2018-04-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (13):
  - Fremont, California
  - Miami, Florida
  - Miramar, Florida
  - Tampa, Florida
  - Arlington Heights, Illinois
  - Carmel, Indiana
  - Fort Gratiot, Michigan
  - Albuquerque, New Mexico
  - New York, New York
  - Stony Brook, New York
  - Dallas, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
- Australia (3):
  - Woolloongabba, Queensland
  - Carlton, Victoria
  - East Melbourne, Victoria
- Canada (2):
  - Hamilton, Ontario
  - Toronto, Ontario
- France (5):
  - Brest
  - Nancy
  - Nice
  - Rouen
  - Thionville
- Germany (11):
  - Augsburg
  - Berlin
  - Bochum
  - Darmstadt
  - Dresden
  - Dülmen
  - Frankfurt
  - Ibbenbueren
  - Lübeck
  - Mahlow
  - Münster
- Rotterdam, Netherlands
- Hamilton, New Zealand
- Gothenburg, Sweden
- United Kingdom (4):
  - Lanarkshire
  - Leeds
  - Manchester
  - Surrey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 42 sites in the USA, Canada, Australia/New Zealand, and Europe from December 2015 to July 2017.
Groups:
- CLS001 (Omiganan) Gel: CLS001 (Omiganan) gel applied once daily
  CLS001 (Omiganan): Topical gel
Period: Double-Blind Study Period
Arm/Group | CLS001 (Omiganan) Gel | Vehicle Gel
Started | 235 | 228
Completed | 211 | 196
Not Completed | 24 | 32
Not completed — Adverse Event | 4 | 9
Not completed — Lost to Follow-up | 2 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 15 | 17
Not completed — Sponsor Decision | 1 | 0
Period: Open-Label Study Period
Arm/Group | CLS001 (Omiganan) Gel | Vehicle Gel
Started | 188 | 175
Completed | 66 | 48
Not Completed | 122 | 127
Not completed — Adverse Event | 10 | 11
Not completed — Lack of Efficacy | 3 | 2
Not completed — Lost to Follow-up | 7 | 8
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 33 | 37
Not completed — Terminated by Sponsor | 66 | 69

BASELINE CHARACTERISTICS:
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Vehicle Gel | Total
Number analyzed (Participants) | 235 | 228 | 463
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 203 | 193 | 396
  >=65 years | 32 | 35 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (13.06) | 51.6 (12.16) | 51 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 137 | 296
  Male | 76 | 91 | 167
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 37 | 80
  Not Hispanic or Latino | 192 | 191 | 383
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 8 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 222 | 221 | 443
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  New Zealand | 6 | 7 | 13
  Canada | 25 | 26 | 51
  Netherlands | 3 | 4 | 7
  Sweden | 10 | 9 | 19
  United States | 81 | 73 | 154
  United Kingdom | 8 | 9 | 17
  Australia | 23 | 21 | 44
  France | 13 | 11 | 24
  Germany | 66 | 68 | 134
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I - Always burn, never tan | 29 | 31 | 60
  II - Usually burn, tans less than average (with difficulty) | 97 | 106 | 203
  III - Sometimes mild burn, tans less than average | 79 | 71 | 150
  IV - Rarely burn, tan more than average (with ease) | 28 | 15 | 43
  V - Rarely burns, tans profusely | 2 | 5 | 7
  VI - Never burns, tans profusely | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Inflammatory Lesion Count From Baseline to Week 12
Description: Change from Baseline to Week 12 in Inflammatory Lesion Count
Time Frame: 12 weeks
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Treatment | Vehicle Gel
Number analyzed (Participants) | 235 | 228
Lesions | -18.1 (1.77) | -13.5 (1.85)
Statistical Analysis 1: Comparison: Treatment vs Vehicle Gel; Test type: Superiority; p = 0.043, ANCOVA

2. Primary Outcome: Percentage of Participants Who Achieved 2 Grade IGA Reduction.
Description: Percentage of participants who achieved 2 grade IGA reduction at Week 12. IGA scores are from 0 to 5 (Clear, Almost Clear, Mild, Moderate and Severe).
Time Frame: 12 weeks
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment | Vehicle Gel
Number analyzed (Participants) | 235 | 228
Percentage of Participants | 26.3 | 16.9
Statistical Analysis 1: Comparison: Treatment vs Vehicle Gel; Test type: Superiority; p = 0.019, Cochran-Mantel-Haenszel

3. Secondary Outcome: Change in the Number of Inflammatory Lesions From Baseline at Week 9
Description: The absolute change in inflammatory lesions from baseline to Week 9
Time Frame: 9 weeks
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Treatment | Vehicle Gel
Number analyzed (Participants) | 235 | 228
Lesions | -17.4 (1.55) | -15.2 (1.60)

4. Secondary Outcome: Change in the Number of Inflammatory Lesions From Baseline at Week 6
Description: The absolute change in inflammatory lesions from baseline to Week 6
Time Frame: 6 weeks
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Treatment | Vehicle Gel
Number analyzed (Participants) | 235 | 228
Lesions | -13.5 (1.44) | -11.8 (1.48)

5. Secondary Outcome: Percentage of Participants Who Achieved 2 Grade IGA Reduction at Week 9.
Description: Percentage of participants who achieved 2 grade IGA reduction at Week 9. IGA scores are from 0 to 5 (Clear, Almost Clear, Mild, Moderate and Severe).
Time Frame: 9 Weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment | Vehicle Gel
Number analyzed (Participants) | 235 | 228
Percentage of Participants | 18.4 | 14.4

6. Secondary Outcome: Percentage of Participants Who Achieved 2 Grade IGA Reduction at Week 6.
Description: Percentage of participants who achieved 2 grade IGA reduction at Week 6. IGA scores are from 0 to 5 (Clear, Almost Clear, Mild, Moderate and Severe).
Time Frame: 6 Weeks
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment | Vehicle Gel
Number analyzed (Participants) | 235 | 228
Percentage of Participants | 13.8 | 8.9

ADVERSE EVENTS:
Time Frame: 12-week in Double-Blind Period and maximum 1 year in Open-Label Period
Groups:
- CLS001 (Omiganan) Gel (Double-Blind Period): CLS001 (Omiganan) topical gel applied once daily for 12-week
- Vehicle Gel (Double-Blind Period): Vehicle topical gel applied once daily for 12-week
- CLS001 (Omiganan) Gel (Open-Label Period): CLS001 (Omiganan) topical gel applied once daily for maximum 1-year
Arm/Group | CLS001 (Omiganan) Gel (Double-Blind Period) | Vehicle Gel (Double-Blind Period) | CLS001 (Omiganan) Gel (Open-Label Period)
All-Cause Mortality (participants affected / at risk) | 0/235 | 0/228 | 0/363
Serious Adverse Events (participants affected / at risk) | 4/235 | 4/228 | 8/363
Other Adverse Events (participants affected / at risk) | 83/235 | 83/228 | 116/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLS001 (Omiganan) Gel (Double-Blind Period) (N=235) | Vehicle Gel (Double-Blind Period) (N=228) | CLS001 (Omiganan) Gel (Open-Label Period) (N=363)
Cholecystitis acute (Hepatobiliary disorders) | 1 (2) | 0 (0) | 1 (1)
Seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Achilles tendon rupture left (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
B-cell non hodgkin lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Acute cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Melanoma in situ of the lentigo maligna type, level 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Herniated vertebral disc (cervical spine) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Primary gonarthrosis left (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Renal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLS001 (Omiganan) Gel (Double-Blind Period) (N=235) | Vehicle Gel (Double-Blind Period) (N=228) | CLS001 (Omiganan) Gel (Open-Label Period) (N=363)
Viral upper respiratory tract infection (Infections and infestations) | 18 (18) | 22 (23) | 41 (57)
Upper respiratory tract infection (Infections and infestations) | 14 (17) | 4 (4) | 13 (15)
Application site dermatitis (General disorders) | 5 (5) | 1 (1) | 5 (5)
Application site pain (General disorders) | 5 (7) | 8 (9) | 6 (6)
Application site pruritus (General disorders) | 5 (5) | 2 (2) | 2 (2)
Application site erythema (General disorders) | 4 (4) | 7 (8) | 5 (6)
Application site dryness (General disorders) | 2 (3) | 5 (5) | 5 (5)
Headache (Nervous system disorders) | 18 (24) | 14 (24) | 19 (27)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 5 (5) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 2 (2)
Rosacea (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (8) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT02547441/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT02547441/SAP_001.pdf